CLINICAL TRIAL: NCT03130010
Title: The Effect of Nefopam on Catheter-related Bladder Discomfort: A Double-blind, Randomized, Controlled, Parallel Design Study
Brief Title: The Effect of Nefopam on Catheter-related Bladder Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-1604/342-006
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2017-04

CONDITIONS: Nefopam; Catheter-related Bladder Discomfort
MeSH Terms: interventions — Nefopam; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Placebo Comparator): One hour before the end of the operation, the control group was received 20 ml of saline.
  Interventions: Drug: Nefopam or saline
- The Nefopam group (Active Comparator): One hour before the end of the operation, the Nefopam group was received 20 mg of nefopam.
  Interventions: Drug: Nefopam or saline

INTERVENTIONS:
Drug: Nefopam or saline — One hour before the end of the operation, the Nefopam group was received 20 mg of nefopam and the saline and the control group was received 20 ml of saline.

SUMMARY:
In the present study, the investigators evaluated whether nefopam 20 mg reduce the catheter-related bladder discomfort in patients undergoing foley catheter insertion

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to insert the catheter a new foley catheter more than 14 Fr in the operation site,
2. Adults 20 to 75years of age
3. American Society of Anesthesiologists Physical Classification 1,2 patients
4. Patients who pre-agreed to the study
5. Male patient

Exclusion Criteria:

1. Neurogenic bladder
2. Patients diagnosed with irritable bladder
3. study drug sensitive or contraindicated
4. Patients with central nervous system or neurological disorder (epilepsy, patients receiving MAO inhibitor)
5. Patients with urethral and prostate disorders
6. Patients with previous history of myocardial infarction
7. Patients with closed angle glaucoma

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
catheter-related bladder discomfort | postoperative 1 hour
  assessment of catheter-related bladder discomfort using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Eunsu Choi, pf, Study Chair — Seoul National Univ. Bundang Hospital
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea